CLINICAL TRIAL: NCT05966441
Title: Evaluating the Effect of Curcumin in Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: Role of Curcumin in Paclitaxel Induced PN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Paclitaxel induced PN
Record Dates: First submitted 2023-04-07; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Paclitaxel; Curcumin; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Curcumin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: * Details of the research steps that the subscriber will be exposed to:
  * Base line evaluation then alignment in either intervention or control group either for taking the interventional drug or standard of care in control group.
  * Blood samples will be collected at baseline.
  * Patient will be given a weekly supply of the medication and will be asked to take his prescribed dose daily.
  * Every week all patients will be asked about their symptoms and if they experience any adverse drug reaction.
  * Patients will receive the interventional drug until the last paclitaxel dose will be taken.
  * After 3 months, another full clinical examination and blood sample will be obtained.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Patients will receive their Paclitaxel-based chemotherapy along with Curcumin at a dose of oral 2g daily till the end of chemotherapy.
  Interventions: Dietary Supplement: Curcumin; Drug: Paclitaxel
- Control group (Placebo Comparator): Patients will receive their Paclitaxel-based chemotherapy only
  Interventions: Dietary Supplement: Curcumin; Drug: Paclitaxel

INTERVENTIONS:
Dietary Supplement: Curcumin — The safety of curcumin has been widely demonstrated, and curcumin has a variety of potential pharmaceutical applications. Curcumin exhibits antioxidant, anti-inflammatory and anticancer properties and has been described as neuroprotective against neurological disorders.
  Many of curcumin's pharmacological benefits arise from its antioxidant or anti-inflammatory properties. Curcumin appears to have significant potential for treatment of diseases that result from oxidative stress.
  Curcumin is provided in soft gelatin capsules each capsule contains 1 g of curcumin and patient is asked to take 2 capsules daily
Drug: Paclitaxel — Paclitaxel (PTX), the most widely used anticancer drug, is applied for the treatment of various types of malignant diseases. Mechanisms of PTX action represent several ways in which PTX affects cellular processes resulting in programmed cell death. PTX is frequently used as the first-line treatment drug in breast cancer Paclitaxel dose in adjuvant therapy after doxorubicin and cyclophosphamide every 3 weeks 175mg/m2 IV or Weekly 80 mg/m2 IV..
  Paclitaxel dose in neoadjuvant therapy every 3 weeks 175 mg/m2 IV.

SUMMARY:
Paclitaxel induced peripheral neuropathy is the most common and serious side effect associated with Paclitaxel treatment in breast cancer patients receiving Paclitaxel.

The efficacy of antioxidant molecules as neuroprotective strategies to preventing the development of peripheral neuropathy has been investigated in preclinical and clinical studies. Vitamin E and Glutathione have been explored as adjuvant therapies to preventing taxane-induced peripheral neuropathy. Other tested neuroprotective treatments with limited success include amifostine, glutamine and acetyl l-carnitine. Curcumin's antioxidant capacity is similar to other potent antioxidants, such as trolox (a vitamin E analog). Curcumin inhibits lipid peroxidation in different tissues, regulates intracellular levels of antioxidant enzymes (e.g., catalase, glutathione peroxidase and superoxide dismutase) and is an effective intracellular reactive oxygen species (ROS) scavenger.

The investigators are going to investigate the neuroprotective effect of Curcumin against Paclitaxel induced peripheral neuropathy.

DETAILED DESCRIPTION:
The work is a prospective, randomized, open label controlled study. A total of 90 breast cancer female patients will be enrolled in the study. Eligible patients will simply be randomized using random allocation generator, after the end of anthracycline adjuvant therapy to one of two groups, Group I: will receive paclitaxel regimen plus 2g of curcumin Group II: will receive paclitaxel regimen only.

The cases involved in the study will be recruited from Ain Shams Teaching Hospital.

All patients presenting to the department were assessed for eligibility according to certain inclusion and exclusion criteria.

Details of the research steps that the subscriber will be exposed to:

* Base line evaluation then alignment in either intervention or control group either for taking the interventional drug or standard of care in control group.
* Blood samples will be collected at baseline.
* Patient will be given a weekly supply of the medication and will be asked to take his prescribed dose daily.
* Every week all patients will be asked about their symptoms and if they experience any adverse drug reaction.
* Patients will receive the interventional drug until the last paclitaxel dose will be taken.
* After 3 months, another full clinical examination and blood sample will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of early stage breast cancer with age > 18 years.
* Performance status of the patients based on Eastern Cooperative Oncology Group (ECOG) from 0 to 2.
* Patients must receive paclitaxel 80 mg/m2 weekly or 175 mg/m2 every 3 weeks for 12 weeks.
* Patients clinical parameters should be (ANC ≥ 1500/mm3). Platelet count 100,000/mm3) (serum total bilirubin < 1.5 mg/dl) and (creatinine < 1.5 mg/dl).

Exclusion Criteria:

* Patients they had any signs and symptoms of clinical neuropathy.
* Diabetes mellitus
* Patients receiving vitamin supplementation including vitamin B1, B6 and B12
* Patients receiving antidepressants, anticoagulants, opioids or anticonvulsants
* Patients had a hypersensitivity to curcumin.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of Curcumin on the incidence and severity of paclitaxel-induced peripheral neuropathy (PIPN) in breast cancer patients. | Baseline
  After each cycle, initial evaluation of response will be done guided by clinical examination and functional assessment and questionnaire.
Evaluate the effect of Curcumin on the damage of nerve fibers induced by paclitaxel. | Baseline
  Nerve growth factor level will be obtained at day 0 and at the end of the paclitaxel course

SECONDARY OUTCOMES:
Evaluate the effect of adding curcumin to paclitaxel-based chemotherapy on response rate in neoadjuvant therapy. | baseline
  CT scan will be done before first dose of paclitaxel and at the end of the course

REFERENCES:
- [Background] Zhang X, Guan Z, Wang X, Sun D, Wang D, Li Y, Pei B, Ye M, Xu J, Yue X. Curcumin Alleviates Oxaliplatin-Induced Peripheral Neuropathic Pain through Inhibiting Oxidative Stress-Mediated Activation of NF-kappaB and Mitigating Inflammation. Biol Pharm Bull. 2020 Feb 1;43(2):348-355. doi: 10.1248/bpb.b19-00862. Epub 2019 Nov 26. PMID 31776306
- [Background] Al Moundhri MS, Al-Salam S, Al Mahrouqee A, Beegam S, Ali BH. The effect of curcumin on oxaliplatin and cisplatin neurotoxicity in rats: some behavioral, biochemical, and histopathological studies. J Med Toxicol. 2013 Mar;9(1):25-33. doi: 10.1007/s13181-012-0239-x. PMID 22648527
- [Background] Babu A, Prasanth KG, Balaji B. Effect of curcumin in mice model of vincristine-induced neuropathy. Pharm Biol. 2015 Jun;53(6):838-48. doi: 10.3109/13880209.2014.943247. Epub 2014 Nov 28. PMID 25429779
- [Background] Saghatelyan T, Tananyan A, Janoyan N, Tadevosyan A, Petrosyan H, Hovhannisyan A, Hayrapetyan L, Arustamyan M, Arnhold J, Rotmann AR, Hovhannisyan A, Panossian A. Efficacy and safety of curcumin in combination with paclitaxel in patients with advanced, metastatic breast cancer: A comparative, randomized, double-blind, placebo-controlled clinical trial. Phytomedicine. 2020 Apr 15;70:153218. doi: 10.1016/j.phymed.2020.153218. Epub 2020 Apr 18. PMID 32335356